CLINICAL TRIAL: NCT01494415
Title: A Phase II Study of Concurrent Nab-Paclitaxel, Carboplatin and Thoracic Radiotherapy in Local Advanced Squamous Cell Lung Cancer
Brief Title: Concurrent Nab-P/Carboplatin and Thoracic Radiotherapy in Squamous Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Shenglin Ma, President of the hospital, First People's Hospital of Hangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZFH CA11-01
Record Dates: First submitted 2011-12-14; First posted 2011-12-19 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell
Keywords: Squamous Cell Lung Cancer; radiation therapy; chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemoradiotherapy (Experimental): This is a single arm study with patients receiving nab-paclitaxel, carboplatin and thoracic radiotherapy.
  Interventions: Drug: Paclitaxel for Injection（Albumin Bound）; Drug: carboplatin; Radiation: thoracic radiation therapy

INTERVENTIONS:
Drug: Paclitaxel for Injection（Albumin Bound） — concurrent: 60 mg/m2, IV, weekly; consolidation: 260 mg/m2, IV, every 3 weeks
  Other Names: Abraxane®
Drug: carboplatin — concurrent: AUC 2, IV, weekly; consolidation: AUC 6, IV, every 3 weeks
Radiation: thoracic radiation therapy — 66 Gy in 33 fractions,both three-dimensional conformal and intensity modulated radiation therapy are allowed

SUMMARY:
Nab-paclitaxel and carboplatin showed better treatment response compared with cremophor-based paclitaxel and carboplatin as first-line therapy in advanced non-small cell lung cancer, especially for squamous cell cancer. The regimen of weekly nab-paclitaxel, carboplatin and concurrent radiotherapy was well tolerated in a phase I study. Given nab-paclitaxel, carboplatin and concurrent radiotherapy in patients with local advanced squamous cell lung cancer may have promising result.

DETAILED DESCRIPTION:
This study was conducted to explore the efficacy and toxicity of concurrent chemoradiotherapy with nab-paclitaxel, carboplatin and thoracic radiotherapy in unresectable local advanced squamous cell lung cancer. Patients will be given nab-paclitaxel weekly at a dose of 60mg/m2, in combination with carboplatin (AUC 2) weekly during concurrent chemoradiotherapy. Thoracic radiation was administered at a dose of 66 Gy/33 fractions, both 3 dimensional conformal and intensity modulated radiation therapy are allowed. Two cycles of consolidation therapy with full dose nab-paclitaxel (260 mg/m2 on day 1) and carboplatin (AUC 6 on day 1) every 21 day will be delivered.

ELIGIBILITY:
Inclusion Criteria:

* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Previously untreated, histological documented, inoperable stage IIIA or IIIB squamous cell carcinoma of lung, excluding those with pericardial, pleural effusion, and those with contralateral hilar or contralateral supraclavicular lymph nodes.
* Patients must have measurable disease according to RECIST criteria, and all detectable tumor can be encompassed by radiation therapy fields.
* Weight loss ≦ 5% in the previous six months.
* Patient must have adequate blood, liver, lungs and kidney function within the requirements of this study.
* Female patients of child-bearing potential must test negative for pregnancy at the time of enrollment based on a serum pregnancy test. Male and female patients must agree to use a reliable method of birth control during and for 3 months following the last dose of study drug.
* Patients must sign a study-specific informed consent form prior to study entry.

Exclusion Criteria:

* Complete tumor resection, recurrent disease, or those patients eligible for definitive surgery.
* Previous chemotherapy or previous biologic response modifiers for current lung cancer.
* Patient has previously had thoracic radiation therapy.
* Prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for five years or more.
* Serious concomitant disorders that would compromise the safety of the patient, or compromise the patient's ability to complete the study, at the discretion of the investigator.
* History of significant neurological or mental disorder, including seizures or dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-07 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
tumor response rate | one month after the end of all treatment

SECONDARY OUTCOMES:
progression-free survival | 2 years from patient enrollment
overall survival | 2 years from patient enrollment
esophagitis | 6 mouths from the initiation of treatment
  acute esophagitis of Grade III and above

CONTACTS AND LOCATIONS:
Overall Officials: Shenglin Ma, MD, Principal Investigator — The First People's Hospital of Hangzhou
Locations (2):
- China (2):
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang